CLINICAL TRIAL: NCT05332132
Title: Evaluation of the Heracure Device for Hysterectomy
Brief Title: Ex Vivo Study of the Heracure Device for Intra-uterine Morcellation After Vaginal or Laparoscopic Hysterectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heracure Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 202019038
Record Dates: First submitted 2022-03-30; First posted 2022-04-18 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-04

CONDITIONS: Vaginal or Laparoscopic Hysterectomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intrauterine Morcellation of Uteri Post-Surgery (Experimental): Intrauterine Morcellation of Uteri Post-Surgery (Ex Vivo Study)
  Interventions: Device: Heracure Device

INTERVENTIONS:
Device: Heracure Device — Intrauterine Morcellation of Uteri Post-Surgery (Ex Vivo Study)

SUMMARY:
Safety and performance evaluation of the Heracure Device for intra-uterine morcellation after vaginal or laparoscopic hysterectomy.

DETAILED DESCRIPTION:
The purpose of this clinical investigation is to evaluate the safety and efficacy of the Heracure Device for intra-uterine morcellation after vaginal or laparoscopic hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

* Subject is undergoing hysterectomy due to benign gynecologic disease

Exclusion Criteria:

* Subject is not suspected of malignancy

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-04-18 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Device or procedure related Adverse Event (AE) | Intra-operation
  Adverse Event defined as uterine perforation at the end of procedure, assessed by inflating the uterus with saline.

SECONDARY OUTCOMES:
Device Success | Intra-operation
  Device Success defined as the ability to reduce uterus size/circumference and the time required for performing the morcellation procedure

CONTACTS AND LOCATIONS:
Overall Officials: Gal Meister, Study Director — Sponsor GmbH
Locations (1):
- Meir Medical Center, Kfar Saba, Israel

REFERENCES:
- [Derived] Pomeranz M, Schonman R, Yagur Y, Tamir Yaniv R, Klein Z, Daykan Y. An intrauterine cavity morcellator: A novel approach to high volume uterus morcellation. Ex-vivo study. PLoS One. 2023 Mar 17;18(3):e0282149. doi: 10.1371/journal.pone.0282149. eCollection 2023. PMID 36930660